CLINICAL TRIAL: NCT01050413
Title: Evaluation of Serum Thymidine Kinase Activity in Diagnosis,Prognosis and Monitoring of Treatment in Patients With Solid Tumors
Brief Title: Evaluation of Thymidine Kinase Activity in the Serum of Patients With Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Tamar Peretz, Head of Oncology Department, Hadassah Medical Organization
Other Study IDs: 044108-HMO-CTL
Record Dates: First submitted 2010-01-05; First posted 2010-01-15 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2009-12

CONDITIONS: Solid Tumors
Keywords: Thymidine Kinase 1 activity; diagnosis; prognosis; follow-up
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: colon cancer, prostate cancer, lung cancer, ovarian cancer

SUMMARY:
This study aimed to evaluate serum thymidine kinase 1 (TK1) activity as a marker for solid tumors and more specifically in: preoperative testing for prediction of disease recurrence and survival; follow-up after surgical removal of the original tumor for early detection of disease recurrence and in monitoring therapy as a surrogate marker of tumor response.

DETAILED DESCRIPTION:
Thymidine kinase 1 (TK1) is a metabolic enzyme catalyzing the ATP-dependent phosphorylation of thymidine to thymidine monophosphate followed by its utilization in DNA synthesis. It has been demonstrated that activity of TK1 in the serum of cancer patients corresponds to the amount of dividing tumor cells. Several clinical investigations clearly showed that abnormal TK1 levels indicate tumor growth. In breast cancer, serum TK1 was shown to predict increased risk of recurrence following surgery and may be a good marker for monitoring the response to therapy. The measurements of TK1 were useful as a prognostic and monitoring factor in patients with NSCLC. Unfortunately, all previously used assays measuring TK1 activity showed relatively low analytical sensitivity. Recently, the novel high sensitive non-radioactive TK1 assay (DiviTum) has been developed. With this assay tumour growth may be detected at an earlier stage of disease and smaller amounts of residual disease may be detected during and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with colon, breast, prostate and lung cancer before and during treatment

Exclusion Criteria:

* pregnant women;
* patients with generalized CMV and HZV infections;
* patients with severe rheumatoid arthritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from oncology department and patients visiting outpatient, daycare oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel